CLINICAL TRIAL: NCT00006094
Title: A Phase I/II Study of Preoperative Oxaliplatin (NSC# 266046), 5-Fluorouracil, and External Beam Radiation Therapy in Locally Advanced Rectal Cancer
Brief Title: Oxaliplatin, Fluorouracil, and External-Beam Radiation Therapy Followed by Surgery in Treating Patients With Locally Advanced Cancer of the Rectum
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02357; CALGB-89901; U10CA031946 (NIH); CDR0000068099 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-08-03; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Rectum; Stage II Rectal Cancer; Stage III Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Fluorouracil

ARMS (1):
- Treatment (oxaliplatin, fluorouracil, EBRT) (Experimental): Patients receive oxaliplatin IV over 1 hour on day 1, fluorouracil IV continuously on days 1-7, and radiotherapy on days 1-5. Treatment repeats weekly for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: oxaliplatin; Drug: fluorouracil; Radiation: external beam radiation therapy

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Radiation: external beam radiation therapy — Undergo external beam radiation therapy
  Other Names: EBRT

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy, radiation therapy, and surgery may be a more effective treatment for cancer of the rectum. Phase II trial to study the effectiveness of combining oxaliplatin, fluorouracil, and external-beam radiation therapy followed by surgery in treating patients who have locally advanced cancer of the rectum

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of oxaliplatin when combined with fluorouracil and external beam radiotherapy in patients with locally advanced adenocarcinoma of the rectum.

(Phase I closed to accrual effective 03/27/2003). II. Determine the pathological response rate in patients treated with this preoperative regimen and surgical resection.

III.Determine the late toxicity of this preoperative regimen in these patients. IV. Determine, in a preliminary manner, the progression-free survival, local control, and overall survival in patients treated with this regimen.

OUTLINE: This is a dose-escalation, multicenter study of oxaliplatin.

Patients receive oxaliplatin IV over 1 hour on day 1, fluorouracil IV continuously on days 1-7, and radiotherapy on days 1-5. Treatment repeats weekly for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of oxaliplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated at that dose level in the phase II portion of the study. (Phase I closed to accrual effective 03/27/2003). Patients may undergo radical resection of rectal tumor within 4-6 weeks after completion of chemoradiotherapy.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 9-24 patients will be accrued for phase I of the study (phase I closed to accrual effective 03/27/2003) and a total of 19 patients will be accrued for phase II of the study within 12-18 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven previously untreated adenocarcinoma of the rectum thatbegins within 12 cm of the anal verge by sigmoidoscopy and/or colonoscopy

  * Locally advanced disease defined as any of the following:

    * Fixed or immovable tumor on physical exam
    * T4 disease with invasion of adjacent structures (e.g., pelvic sidewall, sacral pelvis, bladder, or prostate) by CT scan, rectal ultrasound, or MRI
    * T3 disease with invasion through the wall of the muscularis propria by transrectal ultrasound, CT scan, or MRI
* No distant metastatic disease
* Performance status - ECOG 0-2
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than upper limit of normal (ULN)
* SGOT/SGPT no greater than 2.5 times ULN
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No active second malignancy except nonmelanomatous skin cancer or carcinoma in situ of the cervix
* Patients are not considered to have an active second malignancy if they have completed therapy and are at less than 30% risk of relapse
* No prior or concurrent evidence of neuropathy
* No history of allergy to platinum compounds or antiemetics
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior fluorouracil or platinum-based therapy for any malignancy
* No other concurrent chemotherapy
* Hormonal therapy allowed only for non-disease related conditions (e.g., insulin for diabetes) OR intermittently as an antiemetic (e.g., dexamethasone)
* No prior pelvic irradiation
* No concurrent antiretroviral therapy (HAART) for HIV positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2000-07; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose of oxaliplatin when delivered concurrently with 5-FU and external beam radiation in patients with locally advanced rectal adenocarcinomas | 7 days
Progression-free survival | From protocol entry until documented progression of disease or death from any cause, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method.
Pathological complete response rate | Up to 5 years
  The new regimen will be considered worthy of further investigation if 5 or greater CR's are observed among the 25 patients treated at the MTD. Assuming the new regimen will result in a 30% CR rate, the probability of observing 5 or greater CR's in 25 patients studied is 0.91. For an underlying CR rate of 0.25 this probability is 0.79. The probability of observing 5 or greater CR's if the underlying CR rate is 0.10 is 0.10.
Latent toxicities graded using the Common Toxicity Criteria (CTC) version 2.0 | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David Ryan, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States